CLINICAL TRIAL: NCT01703624
Title: An Investigation of the Efficacy, Tolerability and Safety of a Range of Doses of Orally Inhaled Glycopyrronium Bromide (PSX1002-GB pMDI) in Male and Female Patients With Moderate or Severe Chronic Obstructive Pulmonary Disease
Brief Title: Dose Ranging Study of Glycopyrronium Bromide in Patients With Moderate or Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prosonix Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSX100201; 2012-003791-40 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: glycopyrronium bromide; glycopyrrolate; oral inhalation; COPD; chronic obstructive pulmonary disease; lung function; pharmacokinetics; tolerability; safety; cross-over; single-dose; dose-ranging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- glycopyrronium bromide 12.5mcg (Experimental): glycopyrronium bromide 12.5mcg single dose via pressurised metered dose inhaler (pMDI)
  Interventions: Drug: glycopyrronium bromide
- glycopyrronium bromide 25mcg (Experimental): glycopyrronium bromide 25mcg single dose via pressurised metered dose inhaler (pMDI)
  Interventions: Drug: glycopyrronium bromide
- glycopyrronium bromide 50mcg (Experimental): glycopyrronium bromide 50mcg single dose via pressurised metered dose inhaler (pMDI)
  Interventions: Drug: glycopyrronium bromide
- glycopyrronium bromide 100mcg (Experimental): glycopyrronium bromide 100mcg single dose via pressurised metered dose inhaler (pMDI)
  Interventions: Drug: glycopyrronium bromide
- placebo (Placebo Comparator): placebo single dose via pressurised metered dose inhaler (pMDI)
  Interventions: Drug: glycopyrronium bromide

INTERVENTIONS:
Drug: glycopyrronium bromide — glycopyrronium bromide suspension in HFA
  Other Names: PSX1002-GB

SUMMARY:
This is an investigation of the beneficial effects, tolerability and safety of a range of single doses of orally inhaled glycopyrronium bromide (PSX1002GB pMDI) in male and female patients with moderate or severe chronic obstructive pulmonary disease (COPD). COPD is a long term and progressive disease of the lungs, generally caused by cigarette smoking, but other factors may be involved. Glycopyrronium bromide (GB) appears to be particularly useful in dilating the constricted airways of such patients, with a duration of action variously described as being between 12 and 24 hours.

This study will investigate how well tolerated and safe this medication is at a range of doses. It will also help in the selection of a suitable dose for larger and repeat dose studies, based on measures of lung response. It will also help to determine how often the medication should be given; twice daily, or once daily.

Up to 40 patients will be enrolled into the study, ranging in age from 40 to 75 years of age. Patients will be medically assessed before participation to ensure their suitability. The study will take place in one centre in the UK over five sessions; at each session one dose (2 puffs) of GB or one dose (2 puffs) of placebo will be administered from a simple inhaler device. Neither staff nor patients will know which dose, or if placebo, is being taken. Lung function will be measured for up to 26 hours after the administration of each dose using standard spirometry equipment. Blood samples will be taken over a 24-hour period to check the blood levels of GB. There will be a period of about a week between each dosing session. Patients will be medically reviewed after the study to confirm that no untoward effects are present.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 40-75 years, inclusive
* A clinical diagnosis of moderate to severe COPD (GOLD guidelines)
* Current smokers or ex-smokers with at least 10-pack year smoking history
* Post-bronchodilator FEV1/FVC ratio < 70 % at Screen
* Post-bronchodilator FEV1 ≥ 40 % to < 80 % of predicted at Screen
* Demonstrated to be responsive to ipratropium (defined as at least an 100ml increase in FEV1 following ipratropium 80 µg)
* Ability to perform acceptable spirometry (ATS/ERS guidelines)
* Willing and able to provide written informed consent

Exclusion Criteria:

* Females who are pregnant or lactating at the Screening Visit, or if of childbearing potential not using an acceptable means of birth control throughout the study (defined in protocol)
* Current evidence or recent history of any clinically significant disease (other than COPD) or abnormality in the opinion of the Investigator that would put the subject at risk or which would compromise the quality of the study data (defined in protocol)
* Recent history of hospitalisation due to an exacerbation of airway disease within three months prior to the Screening Visit or randomisation
* Need for increased treatments of COPD within six weeks prior to the Screening Visit or randomisation
* Primary diagnosis of asthma
* Prior lung volume reductions surgery or history of chest/lung irradiation
* Regular use of daily oxygen therapy
* Use of systemic steroids within three months prior to the Screening Visit or during the run-in period
* Respiratory tract infection within six weeks prior to the Screening Visit.
* History of tuberculosis, bronchiectasis or other non-specific pulmonary disease
* History of urinary retention or bladder neck obstructive type symptoms
* History of narrow-angle glaucoma
* Clinically significant abnormal ECG
* Positive Hepatitis B antigen or positive Hepatitis C antibody
* Positive screening test for HIV antibodies
* Current evidence or history of excessive use or abuse of alcohol in the opinion of the Investigator
* Current evidence or history of abusing legal drugs or use of illegal drugs or substances in the opinion of the Investigator
* Donation of 450 ml or more of blood within eight weeks of the Screening Visit
* History of hypersensitivity or intolerance to aerosol medications
* Participation in another investigational drug study where drug was received within 30 days prior to the Screening Visit.
* Inability to comply with study procedures or with study treatment intake, including inability to be trained and/or inability to demonstrate good inhaler technique with Vitalograph AIM

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in one second (FEV1) Area Under the Curve (AUC) | From time zero to 24-hours
  FEV1 time-adjusted AUC(0-24 hours)

SECONDARY OUTCOMES:
Forced Expiratory Volume in one second (FEV1) Area Under the Curve (AUC) | From time zero to 12-hours
  FEV1 time-adjusted AUC(0-12 hours)
Forced Expiratory Volume in one second (FEV1) Area Under the Curve (AUC) | From 12 to 24-hours
  FEV1 time-adjusted AUC(12-24 hours)
Forced Expiratory Volume in one second (FEV1) | From time zero to 24-hours
  Serial FEV1 time-point assessments
Forced Vital Capacity (FVC) Area Under the Curve (AUC) | From time zero to 24-hours
  FVC time-adjusted AUC(0-24 hours), AUC(0-12 hours), AUC(12-24 hours), serial time-point assessment
Forced Expiratory Volume in one second (FEV1) / Forced Vital Capacity (FVC) ratio | From time zero to 24-hours
  Serial FEV1/FVC time-point assessment
Number of subjects reporting adverse events after each treatment as a measure of safety and tolerability | An average of 9 weeks
  Adverse event monitoring will begin once a subject provides informed consent and will continue until study participation is concluded; incidence rates will be summarised by system organ class, preferred term, severity and by reported relationship to study drug for each treatment
Systolic blood pressure | From time zero to 24-hours
  Descriptive statistics will be presented for the serial measurements by treatment
Diastolic blood pressure | From time zero to 24-hours
  Descriptive statistics will be presented for the serial measurements by treatment
Peripheral pulse rate | From time zero to 24-hours
  Descriptive statistics will be presented for the serial measurements by treatment
Electrocardiography (ECG) | From time zero to 24-hours
  Descriptive statistics will be presented for the serial measurements of each of the standard electrocardiographic (12-lead) parameters by treatment
Clinical hematology | An average of 9 weeks
  Clinical hematology measures will be taken at the Screening Visit and at the Safety Follow-up Visit and will consist of: red blood cell count, hemoglobin, hematocrit, mean cell hemoglobin, mean cell hemoglobin concentration, mean cell volume, white blood cell count, differential white blood cell count and platelet count. Data will be summarised using descriptive statistics
Clinical chemistry | An average of 9 weeks
  Clinical chemistry measures will be taken at the Screening Visit and at the Safety Follow-up Visit and will consist of: sodium, potassium, urea, creatinine, uric acid, glucose, calcium, inorganic phosphorus, total bilirubin, alkaline phosphatase, alanine transaminase, aspartate transminase, gamma glutamyl transferase, creatine kinase, total protein, albumin, cholesterol and triglycerides. Data will be summarised using descriptive statistics
Plasma glycopyrronium bromide concentration-time Area Under the Curve (AUC) | From time zero to 24-hours
  AUC (0-infinity) will be extrapolated from serial measures taken over time zero to 24-hours. The descriptive statistics presented by treatment will be: minimum, median, maximum, geometric mean, arithmetic mean and arithmetic standard deviation
Plasma glycopyrronium bromide peak concentration (Cmax) | From time zero to 24-hours
  Cmax will be obtained from serial measures taken over time zero to 24-hours. The descriptive statistics presented by treatment will be: minimum, median, maximum, geometric mean, arithmetic mean and arithmetic standard deviation
Plasma glycopyrronium bromide time to maximum concentration (tmax) | From time zero to 24-hours
  tmax will be calculated from serial measures taken over time zero to 24-hours. The descriptive statistics presented by treatment will be: minimum, median, maximum, geometric mean, arithmetic mean and arithmetic standard deviation
Plasma glycopyrronium bromide concentration elimination half-life (t1/2) | From time zero to 24-hours
  t1/2 will be calculated from serial measures taken over time zero to 24-hours. The descriptive statistics presented by treatment will be: minimum, median, maximum, geometric mean, arithmetic mean and arithmetic standard deviation
Glycopyrronium bromide total plasma clearance following extravascular administration (CL/F) | From time zero to 24-hours
  CL/F will be calculated from serial plasma concentration measures taken over time zero to 24-hours. The descriptive statistics presented by treatment will be: minimum, median, maximum, geometric mean, arithmetic mean and arithmetic standard deviation
Glycopyrronium bromide apparent volume of distribution following extravascular administration (Vz/F) | From time zero to 24-hours
  Vz/F will be calculated from serial plasma concentration measures taken over time zero to 24-hours. The descriptive statistics presented by treatment will be: minimum, median, maximum, geometric mean, arithmetic mean and arithmetic standard deviation

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Down, MB BS FFPM, Study Director — Prosonix Limited, Oxford, UK; Dave Singh, MA MD MRCP, Principal Investigator — Medicines Evaluation Unit, Manchester, UK
Locations (1):
- Medicines Evaluation Unit, Manchester, United Kingdom